CLINICAL TRIAL: NCT01940341
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Tenofovir Alafenamide (TAF) 25 mg QD Versus Tenofovir Disoproxil Fumarate (TDF) 300 mg QD for the Treatment of HBeAg-Negative, Chronic Hepatitis B
Brief Title: Study to Compare Tenofovir Alafenamide (TAF) Versus Tenofovir Disoproxil Fumarate (TDF) in Participants With Chronic Hepatitis B Infection Who Are Negative for Hepatitis B e Antigen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-320-0108; 2013-000626-63 (EudraCT Number)
Record Dates: First submitted 2013-08-20; First posted 2013-09-12 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: HBeAg-negative Chronic Hepatitis B
Keywords: Hepatitis; Tenofovir; Viread
MeSH Terms: conditions — Hepatitis | interventions — tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAF 25 mg (Experimental): TAF + TDF placebo for 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Interventions: Drug: TAF; Drug: TDF Placebo
- TDF 300 mg (Active Comparator): TDF + TAF placebo for 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Interventions: Drug: TDF; Drug: TAF Placebo
- Open-label TAF (Experimental): All participants who complete the double-blind period (96 weeks or 144 weeks) will be eligible to receive open-label TAF until Week 384 of the study.
  After the end of study treatment, participants can either switch to commercially available anti-HBV treatments in their country or will be followed every 4 weeks, for up to 24 weeks off treatment (treatment-free follow-up (TFFU)) for safety assessment.
  Interventions: Drug: TAF

INTERVENTIONS:
Drug: TAF — 25 mg tablet administered orally once daily
  Other Names: Vemlidy®; GS-7340
  Arms: Open-label TAF; TAF 25 mg
Drug: TDF — 300 mg tablet administered orally once daily
  Other Names: Viread®
  Arms: TDF 300 mg
Drug: TAF Placebo — Tablet administered orally once daily
  Arms: TDF 300 mg
Drug: TDF Placebo — Tablet administered orally once daily
  Arms: TAF 25 mg

SUMMARY:
The primary objective of this study is to compare the efficacy, safety, and tolerability of tenofovir alafenamide (TAF) versus tenofovir disoproxil fumarate (TDF) in treatment-naive and treatment-experienced adults with hepatitis B e antigen (HBeAg)-negative chronic hepatitis B virus (HBV) infection.

DETAILED DESCRIPTION:
Study GS-US-320-0108 is a multi-center clinical trial, planned to enroll participants in multiple countries, including China. However, due to the review timeline difference in China, full enrollment was reached in the main study before China was able to participate. Therefore, details for the China cohort was registered separately (NCT02836236) on ClinicalTrials.gov as the China cohort will not be part of the main study analysis.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
* Adult males and non-pregnant, non-lactating females.
* Documented evidence of chronic HBV infection.
* Hepatitis e antigen (HBeAg)-negative, chronic hepatitis B with all of the following:

  * HBeAg-negative and hepatitis B e antibody (HBeAb) positive at screening.
  * Screening HBV DNA ≥ 2 x 10^4 IU/mL.
  * Screening serum alanine aminotransferase (ALT) level > 60 U/L (males) or > 38 U/L (females) and ≤ 10 x the upper limit of the normal range (ULN).
* Treatment-naive participants (defined as < 12 weeks of oral antiviral treatment with any nucleoside or nucleotide analogue), OR treatment-experienced participants (defined as participants meeting all entry criteria [including HBV DNA and serum ALT criteria] and with ≥ 12 weeks of previous treatment with any nucleoside or nucleotide analogue).
* Previous treatment with interferon (pegylated or non pegylated) must have ended at least 6 months prior to Baseline.
* Adequate renal function.
* Normal electrocardiogram (ECG).

Key Exclusion Criteria:

* Females who are breastfeeding.
* Males and females of reproductive potential who are unwilling to use an "effective", protocol-specified method(s) of contraception during the study.
* Co-infection with hepatitis C virus, human immunodeficiency virus (HIV), or hepatitis D virus.
* Evidence of hepatocellular carcinoma.
* Any history of, or current evidence of, clinical hepatic decompensation.
* Abnormal hematological and biochemical parameters, including aspartate aminotransferase (AST) > 10 x ULN
* Received solid organ or bone marrow transplant.
* History of malignancy within the past 5 years, with the exception of specific cancers that are cured by surgical resection; individuals under evaluation for possible malignancy are not eligible.
* Currently receiving therapy with immunomodulators (eg, corticosteroids), investigational agents, nephrotoxic agents, or agents capable of modifying renal excretion.
* Individuals receiving ongoing therapy with drugs not to be used with tenofovir alafenamide or tenofovir disoproxil fumarate or individuals with a known hypersensitivity to study drugs, metabolites, or formulation excipients.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance.
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with dosing requirements.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (105):
- United States (14):
  - Asian Pacific Liver Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Huntington Medical Research Institutes, Pasadena, California
  - Research and Education, Inc., San Diego, California
  - University California San Francisco (UCSF), San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - University of Miami, Miami, Florida
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - ID Care, Hillsborough, New Jersey
  - Sing Chan Private Practice, Flushing, New York
  - New Discovery, LLC, Flushing, New York
  - Xiaoli Ma, PC, Philadelphia, Pennsylvania
  - Hunter Holmes McGuire VA DVMC, Richmond, Virginia
- Australia (5):
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - Zeidler Ledcor Centre Division of Gastroenterology, Edmonton, Alberta
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Dr. John Farley Inc., Vancouver, British Columbia
  - Vancouver Infectious Disease Research and Care Centre, Vancouver, British Columbia
  - Gastrointestinal Research Institute (GIRI), Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- France (2):
  - Hôpital de la Croix Rousse, Lyon
  - Hopital Civil de Strasbourg- CHU Service, Strasbourg
- Hong Kong (4):
  - Queen Mary Hospital, Hong Kong, Hong Kong SAR
  - Princess Margaret Hospital, Kwai Chung
  - Prince of Wales Hospital, Shatin
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
- India (10):
  - Global Hospitals, Hyderabad, Andhra Pradesh
  - Centre for Liver Research & Diagnostic, Deccan College of Medical Sciences and Allied Hospitals, Hyderabad, Andhra Pradesh
  - Nirmal Hospital, Surat, Gujarat
  - Seth GS Medical College and KEM Hospital, Mumbai, Maharashtra
  - Global Hospital Super Specialty & Transplant Centre, Pārel, Mumbai
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - S. R Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Institute of Post Graduate Medical Education And Research, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Institute of Liver and Biliary Sciences, New Delhi
- Italy (4):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera S. Orsola - Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Ospedali, Foggia
  - Azienda Ospedaliero- Universitaria Pisana, Pisa
- Japan (11):
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Kyushu University Hospital Fukuoka, Fukuoka, Fukuoka-shi
  - National Hospital Organization Nagasaki Medical Center, Omura-shi, Nagasaki
  - Osaka University Hospital, Suita, Osaka
  - Shin-Kokura Hospital, Kitakyushu
  - Kobe City Medical Center General Hospital, Kobe
  - Japan Red Cross Musashino Hospital, Musashino
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Osaka Red Cross Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - Medical Hospital of Tokyo Medical and Dental University, Tokyo
- Auckland Clinical Studies Limited, Auckland, New Zealand
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku Klinika, Bialystok
  - Szpital Specjalistyczny w Chorzowie Oddział, Chorzów
  - SPZOZ, Wojewódzki Specjalistyczny Szpital, Lodz
  - Centrum Badan Klinicznych - Przychodnia Badan, Wroclaw
- Romania (5):
  - Institutul National de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest, București
  - Centrul Medical de Diagnostic si Tratament "Dr. Victor Babes", Bucharest
  - Institutul National de Boli Infectioase Prof.Dr. Matei Bals, Bucharest
  - Spitatul Clinic de Boli Infectioase Constanta, Constanța
  - Gastromedica SRL, Iași
- Russia (10):
  - Infection Center LLC Building 20, MSH #163 Territory Koltsovo, Kol'tsovo, Novosibirsk Oblast
  - 1st Moscow State Medical University University Clinical Hospital #3, Moscow
  - Limited Liability Company "Modern Medicine Clinic", Moscow
  - Infectious Clinical Hospital #1 of Moscow Healthcare Department, Moscow
  - Novosibirsk State Medical University, Novosibirsk
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Scientific Research Institute of Clinical Immunology, Novosibirsk
  - Clinical Infectious Hospital named after S.P.Botkin, Saint Petersburg
  - Kirov Medical Military Academy, Saint Petersburg
  - Research Institute of Influenza, Saint Petersburg
- South Korea (10):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yonsei University, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Taiwan (5):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (5):
  - Dicle University Medical Faculty Department of Infectious Diseases, Diyarbakır, Diyarbakri
  - Ankara Üniversitesi Gastroenteroloji Bilim Dalı Cebeci, Ankara
  - Uludag Üniversitesi Tıp Fakültesi Gastroenteroloji, Bursa
  - Istanbul Universitesi Cerrahpassa Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
- United Kingdom (3):
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Barts and The London NHS Trust Royal London Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Derived] Buti M, Lim YS, Chan HLY, Agarwal K, Marcellin P, Brunetto MR, Chuang WL, Janssen HLA, Fung SK, Izumi N, Jablkowski MS, Abdurakhmanov D, Abramov F, Wang H, Botros I, Yee LJ, Mateo R, Flaherty JF, Osinusi A, Pan CQ, Shalimar X, Seto WK, Gane EJ. Eight-year efficacy and safety of tenofovir alafenamide for treatment of chronic hepatitis B virus infection: Final results from two randomised phase 3 trials. Aliment Pharmacol Ther. 2024 Dec;60(11-12):1573-1586. doi: 10.1111/apt.18278. Epub 2024 Sep 27. PMID 39327857
- [Derived] Lim YS, Chan HLY, Ahn SH, Seto WK, Ning Q, Agarwal K, Janssen HLA, Pan CQ, Chuang WL, Izumi N, Fung S, Shalimar, Brunetto M, Hui AJ, Chang TT, Lim SG, Abramov F, Flaherty JF, Wang H, Yee LJ, Kao JH, Gane E, Hou J, Buti M. Tenofovir alafenamide and tenofovir disoproxil fumarate reduce incidence of hepatocellular carcinoma in patients with chronic hepatitis B. JHEP Rep. 2023 Jul 13;5(10):100847. doi: 10.1016/j.jhepr.2023.100847. eCollection 2023 Oct. PMID 37771546
- [Derived] Chan HLY, Buti M, Lim YS, Agarwal K, Marcellin P, Brunetto M, Chuang WL, Janssen HLA, Fung S, Izumi N, Abdurakhmanov D, Jablkowski M, Celen MK, Ma X, Caruntu F, Flaherty JF, Abramov F, Wang H, Camus G, Osinusi A, Pan CQ, Shalimar, Seto WK, Gane E; GS-US-320-0110 and GS-US-320-0108 investigators. Long-Term Treatment With Tenofovir Alafenamide for Chronic Hepatitis B Results in High Rates of Viral Suppression and Favorable Renal and Bone Safety. Am J Gastroenterol. 2024 Mar 1;119(3):486-496. doi: 10.14309/ajg.0000000000002468. Epub 2023 Aug 9. PMID 37561058
- [Derived] Cathcart AL, Chan HL, Bhardwaj N, Liu Y, Marcellin P, Pan CQ, Shalimar, Buti M, Cox S, Parhy B, Zhou E, Martin R, Chang S, Lin L, Flaherty JF, Kitrinos KM, Gaggar A, Izumi N, Lim YS. No Resistance to Tenofovir Alafenamide Detected through 96 Weeks of Treatment in Patients with Chronic Hepatitis B Infection. Antimicrob Agents Chemother. 2018 Sep 24;62(10):e01064-18. doi: 10.1128/AAC.01064-18. Print 2018 Oct. PMID 30038044
- [Derived] Seto WK, Asahina Y, Brown TT, Peng CY, Stanciu C, Abdurakhmanov D, Tabak F, Nguyen TT, Chuang WL, Inokuma T, Ikeda F, Santantonio TA, Habersetzer F, Ramji A, Lau AH, Suri V, Flaherty JF, Wang H, Gaggar A, Subramanian GM, Mukewar S, Brunetto MR, Fung S, Chan HL. Improved Bone Safety of Tenofovir Alafenamide Compared to Tenofovir Disoproxil Fumarate Over 2 Years in Patients With Chronic HBV Infection. Clin Gastroenterol Hepatol. 2018 Jun 20:S1542-3565(18)30633-5. doi: 10.1016/j.cgh.2018.06.023. Online ahead of print. PMID 29933096
- [Derived] Agarwal K, Brunetto M, Seto WK, Lim YS, Fung S, Marcellin P, Ahn SH, Izumi N, Chuang WL, Bae H, Sharma M, Janssen HLA, Pan CQ, Celen MK, Furusyo N, Shalimar D, Yoon KT, Trinh H, Flaherty JF, Gaggar A, Lau AH, Cathcart AL, Lin L, Bhardwaj N, Suri V, Mani Subramanian G, Gane EJ, Buti M, Chan HLY; GS-US-320-0110; GS-US-320-0108 Investigators. 96 weeks treatment of tenofovir alafenamide vs. tenofovir disoproxil fumarate for hepatitis B virus infection. J Hepatol. 2018 Apr;68(4):672-681. doi: 10.1016/j.jhep.2017.11.039. Epub 2018 Jan 17. PMID 29756595
- [Derived] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-320-0108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in East Asia, Europe, North America, Australia, India, and New Zealand.
Pre-assignment Details: 877 participants were screened.
Groups:
- TAF 25 mg: Tenofovir alafenamide (Vemlidy®; TAF) 25 mg + tenofovir disoproxil fumarate (TDF) placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- TDF 300 mg: TDF 300 mg + TAF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- TAF 25 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with Open-label (OL) TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (treatment-free follow-up [TFFU]) for the assessment of safety.
- TDF 300 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to switch to OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
Period: Period 1: Double-blind Phase
Arm/Group | TAF 25 mg | TDF 300 mg | TAF 25 mg to TAF 25 mg | TDF 300 mg to TAF 25 mg
Started | 285 | 141 | 0 | 0
Completed | 261 | 129 | 0 | 0
Not Completed | 24 | 12 | 0 | 0
Not completed — Withdrew Consent | 7 | 4 | 0 | 0
Not completed — Lost to Follow-up | 8 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 0 | 0
Not completed — Investigator's Discretion | 3 | 1 | 0 | 0
Not completed — Non-compliance with Study Drug | 1 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Specified Criteria for Withdrawal | 1 | 0 | 0 | 0
Not completed — Randomized but Never Treated | 0 | 1 | 0 | 0
Period: Period 2: Open-Label TAF Extension Phase
Arm/Group | TAF 25 mg | TDF 300 mg | TAF 25 mg to TAF 25 mg | TDF 300 mg to TAF 25 mg
Started (At the end of Double-blind Phase, participants were given the option to receive TAF in an OL TAF Extension Phase for up to 240 or 288 weeks.) | 0 | 0 | 261 (24 participants from TAF arm did not enter the OL TAF Extension Phase.) | 129 (12 participants from TDF arm did not enter the OL TAF Extension Phase.)
Completed | 0 | 0 | 227 | 118
Not Completed | 0 | 0 | 34 | 11
Not completed — Withdrew Consent | 0 | 0 | 17 | 4
Not completed — Investigator's Discretion | 0 | 0 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 6 | 0
Not completed — Protocol Specified Criteria for Withdrawal | 0 | 0 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — HbsAg Seroconversion | 0 | 0 | 1 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Participants who received at least 1 dose of study drugs.
Groups:
- TAF 25 mg: Double-blind Phase: Tenofovir alafenamide (Vemlidy®; TAF) 25 mg + tenofovir disoproxil fumarate (TDF) placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Open-label TAF extension Phase: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
- TDF 300 mg: Double-blind Phase: TDF 300 mg + TAF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Open-label TAF extension Phase: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
- Total: Total of all reporting groups
Arm/Group | TAF 25 mg | TDF 300 mg | Total
Number analyzed (Participants) | 285 | 140 | 425
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 276 | 136 | 412
  >=65 years | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.6) | 48 (10.4) | 46 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 54 | 166
  Male | 173 | 86 | 259
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 279 | 140 | 419
  Unknown or Not Reported | 4 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 205 | 101 | 306
  Race: White | 71 | 35 | 106
  Race: Black or African American | 5 | 3 | 8
  Race: Other or More Than One Race | 2 | 1 | 3
  Race: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 41 | 28 | 69
  Canada | 29 | 17 | 46
  South Korea | 30 | 15 | 45
  Taiwan | 22 | 15 | 37
  United States | 24 | 13 | 37
  Russia | 22 | 13 | 35
  India | 26 | 7 | 33
  Japan | 21 | 6 | 27
  Romania | 13 | 8 | 21
  Poland | 12 | 6 | 18
  Turkey | 10 | 4 | 14
  New Zealand | 10 | 2 | 12
  Australia | 9 | 1 | 10
  Italy | 6 | 3 | 9
  United Kingdom | 5 | 1 | 6
  France | 2 | 1 | 3
  Spain | 3 | 0 | 3
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 209 | 106 | 315
    CT | 65 | 23 | 88
    TT | 10 | 9 | 19
    Missing | 1 | 2 | 3
HBV DNA [Mean (Standard Deviation); unit: Log10 IU/mL] | 5.7 (1.34) | 5.8 (1.32) | 5.8 (1.33)
Plasma HBV DNA Level [Count of Participants; unit: Participants]
  < 7 log10 IU/mL | 230 | 116 | 346
  ≥ 7 log10 IU/mL - < 8 log10 IU/mL | 42 | 20 | 62
  ≥ 8 log10 IU/mL | 13 | 4 | 17
Oral antiviral (OAV) treatment status [Count of Participants; unit: Participants]
  Treatment Experienced | 60 | 31 | 91
  Treatment Naive | 225 | 109 | 334
Proteinuria by Urinalysis (dipstick) [Count of Participants; unit: Participants] — Urine protein was measured using the dipstick method. Grade 0 = Absent; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe.
  Participants
    Grade 0 | 270 | 135 | 405
    Grade 1 | 13 | 5 | 18
    Grade 2 | 2 | 0 | 2
    Grade 3 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) DNA < 29 IU/mL
Description: The primary efficacy endpoint was determined by the achievement of HBV DNA < 29 IU/mL at Week 48.
Time Frame: Week 48
Population: Full Analysis set: participants who were randomized into the study and received at least 1 dose of study drugs. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: Percentage of participants
Groups:
- TAF 25 mg: TAF 25 mg + TDF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 285 | 140
Percentage of participants | 94.0 | 92.9
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; The null hypothesis was that the TAF group is at least 10% worse than the TDF group with respect to the proportion of participants with HBV DNA < 29 IU/mL at Week 48. The alternative hypothesis was that the TAF group is less than 10% worse than the TDF group with respect to the proportion of participants with HBV DNA < 29 IU/mL at Week 48. Noninferiority was assessed using a 95% confidence interval (CI) approach, with a noninferiority margin of 10%; Test type: Non-Inferiority or Equivalence — Sample sizes of 130 and 260 participants in the TDF group and TAF groups, respectively were planned to give 90% power to rule out the noninferiority margin of 10% at a 1-sided significance level of 0.025. This sample size was based on the assumption that the expected difference (TAF-TDF) in proportion of participants with HBV DNA<29 IU/mL was 0 and the proportion of participants with HBV DNA<29 IU/mL in the TDF group was 91%. All missing data were treated as not achieving the primary endpoint; Difference in proportions = 1.8, 95% CI 2-sided [-3.6 to 7.2] — Difference in the proportion between treatment groups and its 95% CI were calculated based on the Mantel-Haenszel (MH) proportions adjusted by baseline HBV DNA categories and oral antiviral treatment status strata

2. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Hip Dual-Energy X-ray Absorptiometry (DXA) Analysis Set (participants who were randomized, received at least 1 dose of study drugs, and had nonmissing baseline hip BMD values) with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 270 | 133
percentage change | -0.288 (2.1448) | -2.156 (2.1672)

3. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Spine DXA Analysis Set (participants who were randomized, received at least 1 dose of study drugs, and had nonmissing baseline spine BMD values) with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data was excluded from analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 271 | 133
percentage change | -0.876 (2.8558) | -2.514 (3.3558)

4. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data was excluded from analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 275 | 135
mg/dL | 0.01 (0.091) | 0.02 (0.103)

5. Other Pre Specified Outcome: Percentage of Participants With Treatment-emergent Proteinuria by Urinalysis (Dipstick) Through Week 48
Description: Grades 1 (mild), 2 (moderate), and 3 (severe) were the highest treatment-emergent postbaseline grades for urine protein using the dipstick method.
Time Frame: Up to 48 weeks
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 282 | 140
percentage of participants
  Grade 1 | 18.1 | 16.4
  Grade 2 | 1.1 | 2.1
  Grade 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Randomization up to approximately 427.6 weeks Adverse Events: First dose date up to Week 384
Description: All-cause mortality: Randomized Analysis Set: All participants randomized into the study.
  Adverse events: Safety Analysis Set: Participants who received at least 1 dose of study drug in the respective period.
Groups:
- Double-blind Phase: TAF 25 mg: TAF 25 mg + TDF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- Double-blind Phase: TDF 300 mg: TDF 300 mg + TAF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384).
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
- Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to switch to Open-label (OL) TAF 25 mg for additional 288 or 240 weeks (Up to Week 384).
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
Arm/Group | Double-blind Phase: TAF 25 mg | Double-blind Phase: TDF 300 mg | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg
All-Cause Mortality (participants affected / at risk) | 0/285 | 2/141 | 1/261 | 0/129
Serious Adverse Events (participants affected / at risk) | 26/285 | 17/140 | 38/261 | 17/129
Other Adverse Events (participants affected / at risk) | 178/285 | 89/140 | 112/261 | 55/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: TAF 25 mg (N=285) | Double-blind Phase: TDF 300 mg (N=140) | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg (N=261) | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg (N=129)
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Plasmodium vivax infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 6 | 3
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: TAF 25 mg (N=285) | Double-blind Phase: TDF 300 mg (N=140) | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg (N=261) | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg (N=129)
Abdominal pain (Gastrointestinal disorders) | 15 | 3 | 9 | 3
Diarrhoea (Gastrointestinal disorders) | 17 | 5 | 11 | 7
Dyspepsia (Gastrointestinal disorders) | 11 | 8 | 9 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 15 | 2
Nausea (Gastrointestinal disorders) | 18 | 10 | 5 | 1
Fatigue (General disorders) | 17 | 10 | 5 | 4
Influenza (Infections and infestations) | 18 | 9 | 13 | 1
Nasopharyngitis (Infections and infestations) | 40 | 19 | 19 | 10
Pharyngitis (Infections and infestations) | 12 | 4 | 14 | 4
Upper respiratory tract infection (Infections and infestations) | 38 | 16 | 23 | 10
Urinary tract infection (Infections and infestations) | 9 | 8 | 9 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 17 | 16 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 7 | 13 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 7 | 9 | 3
Dizziness (Nervous system disorders) | 8 | 7 | 10 | 4
Headache (Nervous system disorders) | 53 | 15 | 27 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 12 | 13 | 8
Hypertension (Vascular disorders) | 8 | 9 | 15 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years